CLINICAL TRIAL: NCT04730726
Title: In Vivo Multispectral Optoacoustic Imaging of Thyroid Nodules
Acronym: THYNODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Schelto Kruijff, MD PhD, Dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201900301
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with thyroid nodules (Experimental): Patients with thyroid nodules that underwent or will undergo an ultrasound with FNA if indicated and if indicated will be scheduled for a (hemi)thyroidectomy
  Interventions: Device: MSOT Acuity Echo

INTERVENTIONS:
Device: MSOT Acuity Echo — Hybrid optoacoustic and ultrasonography imaging

SUMMARY:
Thyroid nodules are common in clinical practice. Head and neck ultrasound is recommended as a routine examination for all patients with thyroid lesions. The Thyroid Imaging Reporting And Documentation System (TIRADS) criteria helps to estimate the risk of malignancy based on ultrasound patterns and nodule sizes guiding the performance of fine-needle-aspiration (FNA). Approximately 20% of FNA results cannot be specified whether being benign or malig-nant tissue. A definitive diagnosis can only be made from histopathology after diagnostic (hemi)thyroidectomy. However, (hemi)thyroidectomy has disadvantages as it leads to over-treatment and has a risk of postoperative morbidity (e.g. hypothyroidism and laryngeal nerve injury). Furthermore, (hemi)thyroidectomy is known to be associated with poor quality of life. Clearly, there is an unmet need for additional diagnostic tools in order to identify malignant thyroid nodules and thereby support the decision making for treatment of the thyroid.

Multispectral optoacoustic tomography (MSOT) is an innovative, non-invasive imaging method currently available in the UMCG that enables visualization of endogenous chromophores and exogenous contrast agents using the generation of ultrasound waves due to light absorption by using high frequency pulsed laser light. Recently, this system has been used by other groups for non-invasive determination of thyroid nodules. Results show that multispectral optoacoustic imaging of thyroid nodules may distinguish benign from malignant nodules. However, most certainly, a larger cohort is necessary to confirm this finding.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with thyroid nodules who underwent or will undergo an ultrasonography (with TIRADS score) with FNA if indicated and will be scheduled for a (hemi)thyroidectomy if indicated;
2. Age ≥ 18 years;
3. Written informed consent.

Exclusion Criteria:

1. Medical or psychiatric conditions that compromise the patients' ability to give informed consent;
2. Previous surgery in head and neck area
3. Previous radiotherapy in head and neck area
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
MSOT signals of endogenous biomarkers | 2 years
  HbO2, HbR, HbT, sO2, fat, water and collagen

SECONDARY OUTCOMES:
Potential correlation FNA | 2 years
  To explore a potential correlation between endogenous optoacoustic signals in vivo with cytology (the standard-of-care of Bethesda scoring system derived from FNA)
Potential correlation ultrasound | 2 years
  To explore a potential correlation between endogenous optoacoustic signals in vivo with TIRADS ultrasonography scoring system (the scoring system used by radiologists when evaluating the thyroid nodules with ultrasonography).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided